CLINICAL TRIAL: NCT00830583
Title: Pompe Prevalence Study in Patients With Muscle Weakness Without Diagnosis
Acronym: POPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-PP-02
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2009-01

CONDITIONS: Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): pompe's disease suspected patient
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: blood test — There is only a blood test at the beginning.

SUMMARY:
An international consensual group recommends confirming the diagnosis of the Pompe disease after a dried blood spot (DBS) with a dosage of the enzymatic activity in other tissue. This strategy is currently used in the usual practice.

The aim is evaluate the prevalence of the Pompe disease among patients with progressive limb girdle muscular weakness and/or axial deficiency, and/or respiratory insufficiency. The diagnosis will be confirmed using DBS.

DETAILED DESCRIPTION:
In Pompe disease, deficiency of the enzyme acid alpha-glucosidase (GAA) results in accumulation of glycogen within the lyososomes of numerous tissues and cell types especially in muscular cells.

Pompe disease is pan ethnic (but with increased prevalence in the afro-American and Chinese population). Pompe disease is rare with an estimated incidence of 1 in 40,000 births. In France so far, a hundred patients have been diagnosed. The difference of results between the epidemiologic studies published and the number of French patients diagnosed is caused by an under-diagnostic of this pathology, very rare and unknown.

The late onset type of the disease (from childhood to adult) is revealed by progressive muscle weakness generally beginning in proximal muscles of the legs. Respiratory muscle weakness is often the cause of death among patients having respiratory insufficiency.

Recognizing Pompe disease can be challenging, as signs and symptoms may be shared with other disorders (limb girdle muscular dystrophy, dystrophinopathy or inflammatory myopathy).

Muscle biopsies are often used to measure GAA activity and for histology in patients with muscle weakness. But glycogen accumulation in the muscles of patients varies with biopsy site, so the diagnosis of Pompe disease can be missed by using only a muscle biopsy. Fibroblasts can also serve as a source of material for research but cell culture facilities are not easy for clinicians and it takes several weeks to obtain confluent cultures. Then, assays that use blood to diagnose Pompe disease were developed. Therefore, a group of international clinicians and biologists met together in London in December 2006 and established an agreement concerning the various methods of this enzyme dosage. Recently, a test on a DBS (dried blood spot) has been developed. This test is not invasive, easy to collect and transport, requires small sample volume and provides rapid results. This international consensual group recommends confirming the diagnosis of the Pompe disease after a DBS with a dosage of the enzymatic activity in other tissue. This strategy is currently used in the usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years
* The patient and/or the patient's legal representative has given their informed consent in writing before any study procedure is initiated
* Patient with :

Limb girdle muscle weakness or axial weakness And/Or Respiratory insufficiency,With unknown etiology

* Sporadic or familial case compatible with a autosomal recessive disorder
* Patient with muscular biopsy (and specific immunologic analyses) without diagnosis.

Exclusion Criteria:

* Patient with a confirmed and documented diagnosis of an etiologic muscular disease determined by the histological analysis (described in appendix 6) that must have been performed on muscle biopsy.
* Patient familial background known with a X-link or a dominant transmission
* Patient who have had confirmation of a Pompe disease by biochemical analysis and/or by molecular biology
* Patient for whom an GAA enzymatic activity has already been performed and for which the result was normal.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the prevalence of the Pompe disease among patients with progressive limb girdle muscular weakness and/or axial deficiency, and/or respiratory insufficiency. The diagnosis will be confirmed using DBS. | during the first and the only visit

SECONDARY OUTCOMES:
Evaluate the relative sensibility of the diagnosis in the Pompe disease by muscular biopsy with histological methods (PAS and acid phosphatase). | during the first and the only visit
Define the various methods of diagnosis for the Pompe Disease. | during the first and the only visit

CONTACTS AND LOCATIONS:
Overall Officials: Claude Desnuelle, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Claude Desnuelle, Nice, France